CLINICAL TRIAL: NCT05825937
Title: Non-invasive Hemodynamic Monitoring With ClearSight in Patients Undergoing Elective Cardiac or Neurointerventional Surgery: A Prospective Observational Cohort Study
Brief Title: Non-Invasive Blood Pressure Monitoring
Status: Recruiting | Type: Observational
Sponsor: University of Saskatchewan (Other)
Responsible Party: Principal Investigator, Peter Hedlin, Clinical Scientist, Assistant Professor, University of Saskatchewan
Other Study IDs: USask-1795
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-01

CONDITIONS: Blood Pressure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Elective Cardiac Surgery Patients: Patients having elective cardiac surgery, who have given written consent, will have the ClearSight device, along with the standard radial arterial line.
  Interventions: Device: ClearSight System
- Elective Neurointerventional Surgery Patients: Patients having elective neurointerventional surgery, who have given written consent, will have the ClearSight device, along with the standard radial arterial line.
  Interventions: Device: ClearSight System

INTERVENTIONS:
Device: ClearSight System — Patients having either elective cardiac surgery or elective neurointerventional surgery will have blood pressure monitored by the ClearSight device, along with the standard of care radial arterial line, throughout their surgery. The arterial line will be placed on the radial artery contralateral to the upper arm blood pressure cuff. The ClearSight device will then be placed on the third finger of the hand ipsilateral to the radial arterial line.

SUMMARY:
The purpose of this study is to evaluate an alternative way of continuously measuring blood pressure in patients coming for complex surgery. The investigators will directly compare the speed of set up and accuracy of the new ClearSight monitor to those taken by the arterial line monitor, which is the current gold standard for recording blood pressure measurements.

DETAILED DESCRIPTION:
Continuous invasive arterial line monitoring is the most accurate way to monitor a patient's hemodynamics. Being able to rapidly detect a spike or drop in blood pressure is crucial in the care of both surgical and critically ill patients. Major fluctuations in blood pressure have been associated with bleeding, cardiac damage, cognitive dysfunction, stroke, and acute kidney injury. The impact of poor blood pressure control on patient outcomes is influenced not only by how high or low the pressure gets, but how long it remains at those extremes. The alternative to continuous blood pressure monitoring is to use intermittent non-invasive blood pressure cuffs, which typically display a blood pressure measurement every 5 minutes when being used in the operating room. While this might be sufficient for routine, short surgeries and monitoring in stable patients, blood pressure cuffs are inadequate for patients who are unstable or undergoing extensive surgery.

An arterial line monitor involves the insertion of a catheter into the radial artery and allows for the beat by-beat monitoring of blood pressure. The insertion of this monitor is painful, time consuming, and puts the patient at risk of infection, bleeding, nerve injury, and damage to the artery. There are many factors that can complicate the insertion of the arterial line including the presence of peripheral vascular disease, small arteries, large body habitus, and poor patient cooperation. In view of these problems, researchers have investigated non-invasive monitoring systems as alternatives to invasive arterial cannulation, but these data are limited and inconsistent.

A alternative device called the ClearSight monitor, produced by Edwards LifeSciences, provides continuous noninvasive blood pressure monitoring. The ClearSight monitor connects to the patient by wrapping an inflatable cuff around their finger. It will detect the blood volume fluctuations in the finger that occur with each heartbeat. It then converts that volume change data into beat-by-beat hemodynamic information, including blood pressure, mean arterial pressure, cardiac output, stroke volume and stroke volume variation. The ClearSight monitor was developed to advance hemodynamic monitoring of moderate-to high-risk surgery patients, including elderly and obese patients.

Patients receiving elective cardiac or cerebrovascular disease are an ideal population to study. These patients require continuous blood pressure monitoring to prevent radical swings in blood pressure (either high or low), which can put the patient at risk of intracranial hemorrhage and increased intracranial pressure, or tissue ischemia, respectively. In addition, these patients frequently have many comorbid conditions including coronary artery disease, congestive heart failure, peripheral vascular disease, cerebrovascular disease, dementia, chronic obstructive pulmonary disease, hypertension, liver disease, renal disease, obesity, malignancy, and diabetes. Many of these health conditions may compromise and affect ClearSight system's ability to analyze blood pressure. For example, peripheral vascular disease, diabetes, and hypertension can cause arterial damage, arterial stenosis and reduced blood flow to the hands and feet. Consequently, it will be informative to test the ClearSight's accuracy in this medically challenging patient demographic.

The current standard of care for patients coming for elective cardiac or neurointerventional procedures at Royal University Hospital is an invasive arterial cannulation. The purpose of this study is to compare the systolic blood pressure, diastolic blood pressure, and mean arterial blood pressure measured by the non-invasive blood pressure monitor (ClearSight) versus the invasive radial arterial cannulation in these patients.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent
* undergoing elective cardiac surgery OR elective neurointerventional surgery (with standard arterial radial line for continuous blood pressure monitoring)

Exclusion Criteria:

* undergoing emergent cardiac surgery OR emergent neurointerventional surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These participants are receiving either elective cardiac surgery or elective neurointerventional surgery at the Royal University Hospital, Saskatoon.
Sampling Method: Non-Probability Sample
Enrollment: 62 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
systolic blood pressure (SBP), diastolic blood pressure (DBP) and mean arterial pressure (MAP) | duration of surgery
  compare differences in blood pressure parameters (SBP, DBP, MAP) collected by ClearSight system versus gold standard (radial arterial line)

SECONDARY OUTCOMES:
time to place instrument | before surgery
  compare time to place the radial arterial line, and ClearSight finger cuff and wrist strap

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hedlin, PhD MD FRCPC, Principal Investigator — University of Saskatchewan
Locations (1):
- Royal University Hospital, Saskatoon, Saskatchewan, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rogge DE, Nicklas JY, Schon G, Grothe O, Haas SA, Reuter DA, Saugel B. Continuous Noninvasive Arterial Pressure Monitoring in Obese Patients During Bariatric Surgery: An Evaluation of the Vascular Unloading Technique (Clearsight system). Anesth Analg. 2019 Mar;128(3):477-483. doi: 10.1213/ANE.0000000000003943. PMID 30649073
- [Background] Dahan A, Engberts DP, Niesters M. Arterial Line Placement: Safety First. Anesthesiology. 2016 Mar;124(3):528-9. doi: 10.1097/ALN.0000000000000968. No abstract available. PMID 26606174
- [Derived] Goncin U, Liu KK, Rawlyk B, Dalkilic S, Walker MEJ, Norton J, Hedlin P. Comparison of the ClearSight finger cuff monitor versus invasive arterial blood pressure measurement in elective cardiac surgery patients: a prospective observational study. Can J Anaesth. 2024 Nov;71(11):1495-1504. doi: 10.1007/s12630-024-02834-x. Epub 2024 Sep 24. PMID 39317830